CLINICAL TRIAL: NCT02873767
Title: A Subject-Blind, Investigator-Blind, Randomized, Placebo-Controlled, First-In-Human Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Single Ascending Subcutaneous Doses of UCB4019 in Healthy Subjects
Brief Title: A First-In-Human Study With a Single Dose UCB4019 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UP0028; 2016-000772-26 (EudraCT Number)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Healthy Volunteers
Keywords: First in human; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Single dose placebo comparator for each active arm
  Interventions: Other: PL1
- UCB4019 Dose 1 (Experimental): Dose 1 calculated based on body weight
  Interventions: Drug: PR1
- UCB4019 Dose 2 (Experimental): Dose 2 calculated based on body weight
  Interventions: Drug: PR1
- UCB4019 Dose 3 (Experimental): Dose 3 calculated based on body weight
  Interventions: Drug: PR1
- UCB4019 Dose 4 (Experimental): Dose 4 calculated based on body weight
  Interventions: Drug: PR1

INTERVENTIONS:
Drug: PR1 — * Active substance: UCB4019
  * Route of Administration: subcutaneously
  Arms: UCB4019 Dose 1; UCB4019 Dose 2; UCB4019 Dose 3; UCB4019 Dose 4
Other: PL1 — * Active substance: Placebo
  * Concentration: 0.9 % saline
  * Route of Administration: subcutaneously
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and tolerability of single ascending doses of UCB4019 administered by subcutaneous injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Good physical and mental health
* At least 18 and less than 65 years of age
* Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period of 3 months after their last dose of study drug

Exclusion Criteria:

* Total Immunoglobulin G <7 g/L or >16 g/L at the Screening Visit
* Absolute neutrophil count <1.5x10^9/L and/or lymphocyte count <1.0x10^9/L
* Known viral hepatitis, has a positive test for Hepatitis B surface antigen or is Hepatitis C virus antibody positive
* Positive test to Human Immunodeficiency Virus (HIV) 1/2 antibodies
* Past medical history or family history of primary immunodeficiency
* Evidence of latent/active Tuberculosis (TB)
* Active infection or a serious infection within 6 weeks before the first dose of IMP
* Renal impairment
* Hepatic impairment
* Vaccination within 6 weeks before the Screening Visit or intent to have a vaccination before Day 43 of the Safety Follow-up Period
* Subject is splenectomized
* received any IMP or experimental procedure within 90 days before the first dose of IMP
* received UCB7665 in a clinical study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events during the study | Day 1 up to Day 57
  An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Pharmacokinetic samples will be taken predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose and Days 7, 10, 13, 16, 19
Area under the curve from 0 to time t, the time of last quantifiable concentration [(AUC0-t)] | Pharmacokinetic samples will be taken predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose and Days 7, 10, 13, 16, 19
Time to reach Cmax (Tmax) | Pharmacokinetic samples will be taken predose, immediately after the end of infusion, 4, 6, 8, 12, 24, 36, 48, 72, and 96 hours postdose and Days 7, 10, 13, 16, 19
Change from Baseline in total Immunoglobulin G (IgG) concentration at day 7 | Predose (Day 1), Day 7
Change from Baseline in total Immunoglobulin G (IgG) concentration at day 10 | Predose (Day 1), Day 10
Change from Baseline in total Immunoglobulin G (IgG) concentration at day 13 | Predose (Day 1), Day 13

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 887 822 9493)
Locations (1):
- Up0028 001, London, United Kingdom